CLINICAL TRIAL: NCT04760665
Title: Randomized, Superiority, Double Blind Controlled With Placebo, Clinical Trial, to Demonstrate the Effectiveness of Fecal Microbiota Transplantation for Selective Intestinal Decolonization of Patients Colonized by Klebsiella Pneumoniae Carbapenemase (KPC)-Producing
Brief Title: Clinical Trial to Demonstrate the Effectiveness of Fecal Microbiota Transplantation for Selective Intestinal Decolonization of Patients Colonized by Carbapenemase-producing Klebsiella Pneumoniae
Acronym: KAPEDIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of elegible population
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Mikrobiomik Healthcare Company S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAPEDIS
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Carbapenemase-producing Enterobacteriaceae Infection
Keywords: fecal microbiota transplantation; Klebsiella pneumoniae; carbapenemase; intestinal colonization; decolonization
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation (Experimental)
  Interventions: Biological: Fecal microbiota transplantation
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Patients will receive four fecal microbiota transplantation (FMT) capsules. Microbiota is obtained from healthy patients.
  Arms: Fecal microbiota transplantation
Other: Placebo — Patients will receive four oral capsules containing placebo. These capsules will have the same shape, weight and colour as capsules containing FMT.
  Arms: Placebo

SUMMARY:
Infections caused by carbapenemase-producing Enterobacteriaceae are frequent and often associated with high rates of mortality. Colonized patients are at increased risk of infection for these microorganisms. Moreover, they can act as a reservoir facilitating the transmission to other patients. To date, decolonization strategies with antibiotics have not obtained convincing results. For that reason our main objective is to investigate the efficacy of fecal microbiota transplantation (FMT) for selective intestinal decolonization of patients colonized by KPC-producing Klebsiella pneumoniae (Kp-KPC) at 30 days after FMT. Our hypothesis is that FMT is effective and safe for selective intestinal decolonization in patients colonized by Kp-KPC. The design of the study is a randomized, superiority, double blind controlled with placebo clinical trial.

The main variable is the percentage of patients with intestinal decolonization at 30 days after FMT in intention to treat population (all randomized patients). Decolonization will be considered as the abscence of isolation of Kp-KPC in culture from rectal swab together with the abscence of detection of carbapenemase by mean of polymerase chain reaction.

Secondary objectives are:

* To evaluate the safety of FMT.
* To determine if FMT is associated with decrease in the amount of bacteria at 7 days after FMT and 30 days after FMT.
* To evaluate if FMT is associated with persistent intestinal decolonization at 3 months after intervention.
* To study if FMT is associated with decrease in the incidence of Kp-KPC infections at 3 months after intervention.
* To evaluate if FMT is associated with decrease in mortality due to Kp-KPC infections at 3 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age> = 18 years.
* Signature of the informed consent by the patient or legally designated person
* Absence of active infection by carbapenemase-type KPC-producing Klebsiella pneumoniae at the time of assessment as well as in the month prior to inclusion in the study

Exclusion Criteria:

* Terminal situation, or estimated life expectancy of less than 3 months
* Pregnant or lactating women
* Intolerance or inability to take oral medication at the time of assessment
* History of aspiration or dysphagia
* Patients with a history of colectomy, colostomy or ileostomy
* Patients who are receiving or have received antibiotics in the month prior to the inclusion assessment
* Neutrophil count less than 500 cells / mm3
* Anticipation of the use of myelosuppressive treatment (eg. dexamethasone, chemotherapy against to solid tumors or prior to transplantation of hematopoietic progenitories) within 30 days after inclusion in the study
* Hematopoietic stem cell transplantation in the month prior to inclusion in the study
* Presence of clinical signs of mucositis
* Forecast of major abdominal surgical intervention in the month following inclusion in the study
* Patients with a Gianella Score> 12 points
* History of having received decolonization guidelines in the previous 3 months
* Severe food allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Decolonization | 30 days after treatment.
  Percentage of patients with intestinal decolonization after receiving oral capsules of FMT or placebo in intention to treat population.

SECONDARY OUTCOMES:
Percentage of patients with adverse effects | 90 days after treatment.
  Percentage of patients with adverse effects
Bacterial load | 7 days and 30 days after treatment.
  Amount of KPC-producing Klebsiella pneumoniae (Kp-KPC) after intervention
Persistent intestinal decolonization | 90 days after treatment.
  Persistence of intestinal decolonization 90 days after intervention
Infections caused by Kp-KPC | 90 days after treatment.
  Percentage of patients with infections caused by Kp-KPC after intervention
Mortality | 90 days after treatment.
  Percentage of patients died after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Castón Osorio, MD, Principal Investigator — Hospital Universitario Reina Sofía; Ángela Cano Yuste, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publishing the results in a journal.
Access Criteria: Upon request to uicec@imibic.org

REFERENCES:
- [Derived] Perez-Nadales E, Cano A, Recio M, Artacho MJ, Guzman-Puche J, Doblas A, Vidal E, Natera C, Martinez-Martinez L, Torre-Cisneros J, Caston JJ. Randomised, double-blind, placebo-controlled, phase 2, superiority trial to demonstrate the effectiveness of faecal microbiota transplantation for selective intestinal decolonisation of patients colonised by carbapenemase-producing Klebsiella pneumoniae (KAPEDIS). BMJ Open. 2022 Apr 6;12(4):e058124. doi: 10.1136/bmjopen-2021-058124. PMID 35387830